CLINICAL TRIAL: NCT03076632
Title: Acute Interactions Between Electromagnetic Stimulation and Physical Exercise
Brief Title: Interactions Between Neurostimulation and Physical Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding obtained to conduct expanded study - to be posted to ClinicalTrials.gov.
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Noam Y. Harel, MD, PhD, Staff Physician, Bronx VA Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: HAR-16-042
Record Dates: First submitted 2017-02-23; First posted 2017-03-10 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Spinal Cord Injuries; Amyotrophic Lateral Sclerosis
Keywords: transcranial magnetic stimulation; neurostimulation; non-invasive stimulation; closed-loop stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Each subject will receive combinations of brain stimulation, cervical stimulation, or peripheral nerve stimulation, either with or without performing simultaneous hand exercises.
Who Masked: Outcomes Assessor
Masking Description: Raw electromyography data assessed while masked to specific conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-disabled volunteers (Active Comparator): Volunteers without neurological injury.
  Interventions:
  * Cervical plus transcranial stimulation
  * Cervical stimulation plus hand/wrist exercise
  * Electromyographic (EMG)-triggered (closed-loop) stimulation
  Interventions: Device: Cervical plus transcranial stimulation; Device: Cervical stimulation plus hand/wrist exercise; Device: Electromyographic (EMG)-triggered (closed-loop) stimulation
- Spinal cord injury (Active Comparator): Volunteers with motor-incomplete cervical spinal cord injury.
  Interventions:
  * Cervical plus transcranial stimulation
  * Cervical stimulation plus hand/wrist exercise
  * Electromyographic (EMG)-triggered (closed-loop) stimulation
  Interventions: Device: Cervical plus transcranial stimulation; Device: Cervical stimulation plus hand/wrist exercise; Device: Electromyographic (EMG)-triggered (closed-loop) stimulation
- Amyotrophic lateral sclerosis (Active Comparator): Volunteers with amyotrophic lateral sclerosis.
  Interventions:
  * Cervical plus transcranial stimulation
  * Cervical stimulation plus hand/wrist exercise
  * Electromyographic (EMG)-triggered (closed-loop) stimulation
  Interventions: Device: Cervical plus transcranial stimulation; Device: Cervical stimulation plus hand/wrist exercise; Device: Electromyographic (EMG)-triggered (closed-loop) stimulation

INTERVENTIONS:
Device: Cervical plus transcranial stimulation — Conditioning pulses of cervical electrical stimulation will be delivered before or after test pulses of transcranial magnetic stimulation.
Device: Cervical stimulation plus hand/wrist exercise — Pulses of cervical stimulation will be delivered while the subject performs finger and wrist motor tasks.
Device: Electromyographic (EMG)-triggered (closed-loop) stimulation — Force and EMG activity of specific hand muscles will be used to trigger peripheral nerve electrical stimulation or transcranial magnetic stimulation.

SUMMARY:
* People with cervical spinal cord injury (SCI) and amyotrophic lateral sclerosis (ALS) have reduced connections in the nerve circuits between the brain and the hands. Activating spared nerve circuits is one potential way to improve recovery.
* The investigators are testing different combinations of physical wrist and hand movements paired with magnetic brain stimulation and electrical spinal cord or nerve stimulation to see the effects on nerve transmission to hand muscles.
* This is a preliminary study. This study is testing for temporary changes in nerve transmission to hand muscles. There is no expectation of long-term benefit from this study. If temporary changes are seen in this study, then future studies would focus on how to prolong that effect.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) and amyotrophic lateral sclerosis (ALS) result in a mixture of destroyed, damaged, and spared neural circuits. Activating spared nerve circuits augments neural transmission.

With this goal in mind, the investigators recently developed a novel method of cervical electrical stimulation (CES) to noninvasively activate arm and hand muscles. The investigators are conducting a pilot clinical study (NCT02469675) to establish CES safety in subjects with cervical SCI, ALS, and non-disabled volunteers. To date, 19 subjects have undergone >120 CES sessions without major safety or tolerability issues.

The current study is designed to gain further mechanistic insight. In Aim 1, the investigators will test in more detail how CES (traveling through spinal and peripheral circuits) interacts with individual pulses of TMS (traveling through corticospinal circuits). In Aim 2, the investigators will further test CES's therapeutic potential by combining stimulation with simultaneous physical exercises. In Aim 3, the investigators will compare the acute effects on synaptic transmission of passive stimulation to stimulation triggered by the subject's own muscle activity.

Please note, this is a preliminary study. This study is testing for temporary changes in nerve transmission to hand muscles. There is no expectation of long-term benefit from this study. If the investigators see temporary changes in this study, then future studies would focus on how to prolong that effect.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 and 65 years;
2. Chronic (more than 12 months since injury) incomplete SCI between levels C2-C8 or diagnosis of definite or probable ALS;
3. Incomplete weakness of left or right hand muscles: score of 2, 3, or 4 (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction;
4. Detectable F-wave responses of the left or right abductor pollicis brevis muscle to median nerve stimulation.

Exclusion Criteria:

1. Multiple spinal cord lesions;
2. History of seizures;
3. Ventilator dependence or patent tracheostomy site;
4. Use of medications that significantly lower seizure threshold, such as tricyclic antidepressants, amphetamines, neuroleptics, dalfampridine, and bupropion;
5. History of stroke, brain tumor, brain abscess, or multiple sclerosis;
6. History of moderate or severe head trauma (loss of consciousness for greater than one hour or evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging);
7. History of implanted brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants, or cardiac pacemaker/defibrillator;
8. Significant coronary artery or cardiac conduction disease;
9. Recent history (within past 6 months) of recurrent autonomic dysreflexia, defined as a syndrome of sudden rise in systolic pressure greater than 20 mm Hg or diastolic pressure greater than 10 mm Hg, without rise in heart rate, accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, and blurry vision (this will be closely monitored during all screening and testing procedures);
10. History of bipolar disorder;
11. History of suicide attempt;
12. Active psychosis;
13. Heavy alcohol consumption (greater than equivalent of 5 oz of liquor) within previous 48 hours;
14. Open skin lesions over the face, neck, shoulders, or arms;
15. Pregnancy
16. Unsuitable for study participation as determined by study physician.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potentials (MEP) | Four visits (3 for non-disabled volunteers) taking place over 2 to 6 weeks.
  Change in MEP amplitude of hand and wrist muscles in response to conditioned versus unconditioned pulses of TMS
Volitional electromyographic (EMG) activity | Four visits (3 for non-disabled volunteers) taking place over 2 to 6 weeks.
  Change in EMG activity of hand and wrist muscles in response to cervical stimulation during physical activity
Response to closed-loop stimulation | Four visits (3 for non-disabled volunteers) taking place over 2 to 6 weeks.
  Transmission of pulses of TMS or peripheral nerve stimulation will be increased when stimulation is triggered by endogenous EMG activity.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y. Harel, MD, PhD, Principal Investigator — James J. Peters VAMC

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.